CLINICAL TRIAL: NCT00419549
Title: Effect of Transdermal Glyceryl-Trinitrate and Parecoxib (Valdecoxib) for the Prevention of Post -ERCP Pancreatitis
Brief Title: Efficacy Study of Glyceryl-Trinitrate Patch and Parecoxib (Valdecoxib) for the Prevention of Pancreatitis After Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Because one of the drugs Valdecoxib was withdrawn due to safety concerns.
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Pramod Kumar Garg, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GE-ERCP-AP/2006
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: ERCP; Pancreatitis
Keywords: ERCP; Pancreatitis; Nitroglycerine; Valdecoxib
MeSH Terms: conditions — Pancreatitis | interventions — Nitroglycerin; valdecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Valdecoxib
  Interventions: Drug: Valdecoxib
- 2 (Active Comparator)
  Interventions: Drug: Glyceryl - trinitrate
- 3 (No Intervention)

INTERVENTIONS:
Drug: Glyceryl - trinitrate — Transdermal Patch once only
  Arms: 2
Drug: Valdecoxib — Single parenteral administration
  Arms: 1

SUMMARY:
ERCP is a diagnostic and therapeutic procedure that is required in patients with suspected common bile duct stone, malignant biliary obstruction, biliary fistula, etc. Pancreatitis may occur as a complication of this procedure after about 5-10% of the ERCP procedures. This complication manifests as persisting pain 24 hours or more after ERCP, along with raised levels of pancreatic enzymes in the blood. Most of the cases of post-ERCP pancreatitis are mild, but may be severe and lead to prolonged hospitalization a few patients. The occurrence of this complication is unpredictable. There have been a number of attempts to prevent this complication. These include giving certain drugs before ERCP e.g. octreotide, somatostatin, steroids, etc. However, these have not been successful. Recently, a study showed that application of glyceryl trinitrate patch on the skin before ERCP might reduce the incidence of post ERCP-pancreatitis. Another study showed that per rectal administration of diclofenac tablet after the ERCP procedure also reduced occurrence of post ERCP pancreatitis. Other experimental studies have shown that certain anti-inflammatory drugs like cox-2 inhibitors may also be effective.

The investigators want to study whether transdermal patch of glyceryl trinitrate or administration of injectable cox-2 inhibitor Valdecoxib (pro-drug Parecoxib) can prevent post-ERCP pancreatitis in our patients who undergo an ERCP.

DETAILED DESCRIPTION:
Acute pancreatitis represents the most common complication after ERCP. The reported incidence of this complication varies from less than 1% to 40%, but rates of about 10% are reported in most prospective studies involving non-selected patients. Although most episodes (about 90%) of post-ERCP pancreatitis are mild, a small percentage of patients (about 10%) may develop severe pancreatitis resulting in significant morbidity and occasional mortality. Despite technical improvements in recent years, the incidence of this complication has not decreased.

The risk factors for development of post ERCP acute pancreatitis are now well known. Balloon dilatation of sphincter of Oddi, difficult papillary cannulation, pancreatic sphincterotomy and multiple pancreatic duct injections have been found to be independent risk factors for post-procedure pancreatitis (Odds ratio of 4.5, 3.4, 3.1, 2.7 respectively) in a recent prospective, multicenter study by Freeman et al. Opacification of the main pancreatic duct alone (MPD) is associated with a 31% incidence of hyperamylasemia. This figure is similar to the 24% incidence of hyperamylasemia which occurs after cholangiography alone. However both injection pressure and volume of contrast medium injected into the pancreatic duct contribute to ductal epithelial or acinar injury by disruption of the intercellular tight junctions with a backflow into the interstitial space.

The role of the osmolarity and ionic nature of the contrast medium is controversial. However non-ionic, low osmolarity contrast media is preferred by most endoscopists. Electrocautery in the vicinity of the MPD orifice may produce edema of the tissues with subsequent obstruction. Etta et al recently showed that use of pure cutting current significantly reduced pancreatitis rates when compared with blended current (3% vs 11%).Precut or access papillotomy is associated with higher risk of pancreatitis when used by endoscopists with less experience, but not in the hands of experienced endoscopists.Operator experience also seems to be a potential risk factor for post ERCP complications. Large volume centers performing > 200 procedures per year had significantly less overall complications (2.0% vs 7.1%, p<0.001) and less complication related deaths (0.18% vs 0.75%, p<0.05), compared to low volume centers in a large Italian multicenter prospective study.

Various agents have been tried with an aim to prevent post ERCP pancreatitis in the last 10 years. These include Gabexate, Somatostatin, Nifedipine, Octreotide, Hydrocortisone, Prednisone, Allopurinol, Interleukin-10, and Methylprednisolone which have been evaluated in randomized controlled studies.Of these agents only Interleukin-10, Somatostatin and Gabexate have been found efficacious. However 13 patients need to be treated prophylactically with Somatostatin and 27 with Gabexate to prevent a single case of post ERCP pancreatitis. Hence these agents are unlikely to be cost-effective or universally applicable. The ideal agent to prevent this complication should be cheap, widely applicable and have a rational basis.

It has been found that cannulation trauma to the papilla or electrocautery leads to sphincter of Oddi spasm and/or papillary edema, thus obstructing free flow of pancreatic juice and contrast with resultant acute pancreatic inflammation.

Akashi et al recently showed that although the frequency of pancreatitis was higher in patients who underwent sphincterotomy, the frequency of severe pancreatitis within 48 hours and the worsening of pancreatitis after 48 hours is significantly lower in this group. Thus the lowering of intraductal pressure after endoscopic sphincterotomy (ES) mitigates the severity of post procedural pancreatitis.

In fact pancreatic stent placement has been shown to be effective for the prevention of post ERCP pancreatitis in high risk patients. In a recent randomized trial, patients had either a 5 Fr nasopancreatic catheter/a stent placed at the end of ERCP or no endoprosthesis was placed. Patients undergoing MPD stenting had a lower frequency of pancreatitis as compared with those in the control group (28% vs 5%, p<0.05)10 However pancreatic stenting on a regular basis is difficult and impractical solution. Repeated attempts to place the pancreatic stent may cause more harm, and a second procedure may be required to remove the stent. Hence instituting adequate drainage of MPD at the end of ERCP seems to be rational and useful but pharmacological rather than mechanical means may be desirable.

Sphincter of Oddi relaxation is modified by cholecystokinin (CCK), vasoactive intestinal peptide (VIP) and nitric oxide (NO) in the physiological state besides a complex neural control involving sympathetic, parasympathetic and enteric nervous system. Jurkowska et al studied the role of nitric oxide (NO) in cerulein induced rat pancreatitis model. It was found that glyceryl trinitrate (NTG, a NO donor) and L-arginine (a substrate for NO synthesis) resulted in significant attenuation of pancreatic damage as well as earlier recovery and augmented cell proliferation in comparison to the saline treated or L-NNA (NO synthase inhibitor) group.

In a randomized double-blind study, prophylactive treatment with NTG (2mg given sublingually 5 min before endoscopy) was compared with placebo in 186 patients. The incidence of pancreatitis was lower in the NTG group compared with placebo (7 of 90 vs 17 of 96; p<0.05). Mean serum amylase values were similar in the two groups.

A more recent study tested the hypothesis that transdermal NTG could be effective in the prevention of post ERCP pancreatitis. One hundred forty-four patients were randomized: 71 received a 15mg NTG patch and 73 a placebo patch. In the control group pancreatitis developed in 11 patients versus 3 in the NTG group (p<0.05). Twenty four hour to baseline serum amylase and lipase ratios were also lower in the NTG group. Hence NO donors seem efficacious in preventing hyperamylasemia and post ERCP pancreatitis Regardless of the initial trigger, the acinar cell injury leads to oxidative stress, nuclear translocation of nuclear factor kappa-B and subsequent transcription of chemo and pro-inflammatory cytokines. This is followed by chemo-attraction and activation of macrophages, T lymphocytes and neutrophils, which are responsible for acinar necrosis and amplification of the pro-inflammatory cascade. Finally after amplification by Kupffer cells, systemic inflammatory response syndrome and multiple organ dysfunction occur. All these events occur within a very short period of time, likely within an hour or two. There is thus a very short therapeutic window during which it is theoretically possible to shut the inflammatory cascade.

Cyclooxygenases (COX) are key enzymes of prostaglandin synthesis and have important role in the regulation of inflammation. Both isoforms of COX are synthesized in acinar cells and their expression is differentially regulated. Upon induction of pancreatitis in the rat model, COX-2 mRNA increases while COX-1 expression remains constant. Song et al studied the effect of pharmacological inhibition of COX-2 and genetic deletion of COX-2 in cerulein induced acute pancreatitis in mice. In both groups, the severity of pancreatitis and pancreatitis induced lung injury was reduced compared with the non-inhibited strains of COX-2 sufficient mice. This indicates that COX-2 plays an important proinflammatory role in pancreatitis and that COX-2 inhibitors may be beneficial in preventing acute pancreatitis or reducing its severity.

Parecoxib is the prodrug of Valdecoxib -a selective COX-2 inhibitor. Following IV or IM injection, Parecoxib is rapidly converted to Valdecoxib, the pharmacologically active substance by enzymatic hydrolysis in the liver. Following a single intramuscular injection of 20mg of Valdecoxib, peak blood levels are achieved in approximately 1 hour. Parecoxib demonstrates an incidence of gastroduodenal ulceration similar to placebo and in twice daily doses had no effect on platelet aggregation or bleeding compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and above undergoing first ERCP procedure

Exclusion Criteria:

* Active acute pancreatitis,
* Lower end malignant bile duct block,
* Patients undergoing repeat procedures,including those with previous sphincterotomy
* Ongoing therapy with nitrates, calcium channel blockers, somatostatin or octreotide
* Patients with bleeding diathesis.
* Patients with chronic pancreatitis
* Patients with cardiac comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2003-10; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Frequency of acute pancreatitis after ERCP | 48 hours

SECONDARY OUTCOMES:
Frequency of pain | 24 hours
Degree of hyper-amylasemia | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pramod K Garg, M.D., D.M., Study Director — All India Institute of Medical Sciences; Vikram Bhatia, M.D., D.M., Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, India

REFERENCES:
- [Background] Kaffes AJ, Bourke MJ, Ding S, Alrubaie A, Kwan V, Williams SJ. A prospective, randomized, placebo-controlled trial of transdermal glyceryl trinitrate in ERCP: effects on technical success and post-ERCP pancreatitis. Gastrointest Endosc. 2006 Sep;64(3):351-7. doi: 10.1016/j.gie.2005.11.060. Epub 2006 May 19. PMID 16923481
- [Background] Moreto M, Zaballa M, Casado I, Merino O, Rueda M, Ramirez K, Urcelay R, Baranda A. Transdermal glyceryl trinitrate for prevention of post-ERCP pancreatitis: A randomized double-blind trial. Gastrointest Endosc. 2003 Jan;57(1):1-7. doi: 10.1067/mge.2003.29. PMID 12518122
- [Background] Cheng CL, Sherman S, Watkins JL, Barnett J, Freeman M, Geenen J, Ryan M, Parker H, Frakes JT, Fogel EL, Silverman WB, Dua KS, Aliperti G, Yakshe P, Uzer M, Jones W, Goff J, Lazzell-Pannell L, Rashdan A, Temkit M, Lehman GA. Risk factors for post-ERCP pancreatitis: a prospective multicenter study. Am J Gastroenterol. 2006 Jan;101(1):139-47. doi: 10.1111/j.1572-0241.2006.00380.x. PMID 16405547
- [Background] Freeman ML, Guda NM. Prevention of post-ERCP pancreatitis: a comprehensive review. Gastrointest Endosc. 2004 Jun;59(7):845-64. doi: 10.1016/s0016-5107(04)00353-0. No abstract available. PMID 15173799
- See also: Patient information database with comprehensive details of ERCP and its complications, including pancreatitis — http://patients.uptodate.com/topic.asp?file=biliaryt/10141